CLINICAL TRIAL: NCT06270355
Title: Stockholm Mammography Risk Stratified Trial
Acronym: SMART
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Hall, Professor, PhD, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023-06555-01
Record Dates: First submitted 2023-12-19; First posted 2024-02-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Women randomised to the experimental arm / individualised screening will have their 2-year breast cancer risk assessed upfront. This is done via an AI (artificial intelligence) derived analyses of the mammograms. Women scored with the highest 2-year risk will be offered a contrast enhanced mammography and an additional mammography at 12 months.
  Interventions: Procedure: Risk based screening
- No intervention arm (Active Comparator): The 35,000 women randomised to the no intervention arm will continue in the Swedish National Breast Cancer Screening Program. This means that they are invited for the next mammography screening after 24 months.
  Interventions: Procedure: Risk based screening

INTERVENTIONS:
Procedure: Risk based screening — Women randomised to the individualised screening arm and judged to be at high risk will be invited to a contrast enhanced mammography and a mammography after 12 months. The intervention is thus a different selection of women compared to what is done today.

SUMMARY:
SMART is a Phase III, randomised, non-blinded screening trial. Women who consent to participate in SMART are randomised to either individualised screening or screening according to the Swedish National Breast Cancer Screening Program. Women randomised to individualised screening get their 2-year risk of breast cancer assessed and women with the highest short-term risk are offered contrast enhanced mammography and a mammogram at 12 months.

DETAILED DESCRIPTION:
Aims: The overarching aim of SMART is to compare the effectiveness of current screening practice with individualised breast cancer screening. In SMART women who recently had a normal mammogram will be randomised to either age based or individualised screening. Women randomised to individualised screening will have their 2-year breast cancer risk assessed upfront. This is done via an artificial intelligence (AI) derived analyses of the mammograms. Women scored with the highest 2-year risk will be offered a contrast enhanced mammography and an additional mammography at 12 months. The possible benefits of individualised screening will be contrasted to the possible harms defined as unnecessary recalls, biopsies and induced anxiety and worry.

Primary Objectives: The primary benefit endpoint is a comparison of the proportion of interval cancers in the intervention and comparison group. The primary safety endpoint is the number of screen-initiated recalls and biopsies which do not lead to a cancer diagnosis.

Secondary Objectives: The secondary benefit endpoint is a comparison of the tumor characteristics of diagnosed cancers in the intervention and comparison group. The investigators will also compare differences in cancer worry, anxiety and / or depression between the intervention and control groups.

Explorative Objectives: To describe the possible side effects related to contrast enhanced mammography and compare them to those experienced after an ordinary mammogram. Cost-effectiveness as measured using incremental cost-effectiveness ratio and willingness-to-pay amount.

Primary Endpoint: For women at high 2-year risk in the intervention arm interval cancers are defined as cancers diagnosed in the interval between contrast enhanced mammography (CEM) and 12-month mammogram plus in the interval between 12- and 24-month interval. For the remaining women in the trial interval cancers are defined as cancers diagnosed between baseline mammography and 24-month mammography.

Information on date of diagnosis and mode of detection (screen detected or interval cancer) is derived from the National Quality Registry for Breast Cancer. To certify the correct diagnosis, the investigators will also use the electronic medical records, Take Care, at Södersjukhuset. Information on number of recalled women and number of biopsies will gathered from the Radiation Information System at the hospital.

Secondary Endpoint: Information on date of diagnosis and tumour characteristics (eg. stage, receptor status) is derived from the National Quality Registry for Breast Cancer. The investigators will compare how the screening modalities are perceived using answers from the self-reported Cancer Worry Scale and State Trait Anxiety Inventory.

Explorative Endpoint: The possible side effects related to contrast enhanced mammography and ordinary mammography will be identified using the self-reported Test Morbidity Index.

Study design: SMART is a Phase III, randomised, non-blinded screening trial. Women who consent to participate in SMART are randomised to either individualised screening or screening according to the Swedish National Breast Cancer Screening Program. Women randomised to individualised screening get their 2-year risk of breast cancer assessed and women with the highest short-term risk are offered contrast enhanced mammography and a mammogram at 12 months.

Study population: Women invited for screening according to the Swedish National Breast Cancer Screening Program at Södersjukhuset, that is, age range 40 - 74 years of age, will be invited to participate in SMART.

Number of included participants: Participants will be matched 1:1 with 35,000 women in each arm.

Intervention: Women randomised to the individualised screening arm and judged to be at high risk will be invited to a contrast enhanced mammography and a mammography after 12 months. The intervention is thus a different selection of women compared to what is done today.

Study Duration: There will be two database locks in SMART. The primary lock is done after approximately four years and two months. Women participating in SMART are part of the initial recruitment phase for a total of two years. They perform mammograms at baseline and 24 months. Adding the 2 year follow up for the lastly recruited participant makes a full trial period 4 years in total, with a further two months allowed to capture women whose scan is delayed. After two months the investigators will consider that screening visit to have been missed. The number of high-risk women will be slightly more than 6,000 in each arm (see 10.1 Population / Power). In addition, a second data lock will be performed after 8 years and two months from the start of the trial, that is, after a fourth round of screens (baseline plus 3 routine follow up mammograms). The same objectives and endpoints will be addressed as after the first data base lock with the exception of questionnaire data. Questionnaire data will only be collected between baseline and the next screen in 24 months. SMART will start in 2024, recruit women for 2 years and follow all women for 6 years. The study will thus end in 2032.

ELIGIBILITY:
Inclusion Criteria:

* Have read, understood and signed the informed consent
* Perform breast cancer screening at Södersjukhuset
* Females in the age range 40 - 74 years at baseline mammography
* Using a smartphone or tablet with BankID

Exclusion Criteria:

* Pregnant, breast feeding or planning to become pregnant.
* Previous breast cancer
* A medical condition that according to the responsible physician would negatively affect the health of the women.
* Cognitive impairment and / or language ability that would make it difficult for the participant to understand the implication of study and to perform a contrast mammography.

For women that will be offered contrast enhanced mammography the clinically accepted and applied exclusion criteria will be used. Women who cannot perform a contrast mammography will be offered an automated ultrasound.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Registered as a woman in the Swedish social security number system.
Enrollment: 70000 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2028-04-08 (Estimated); Study Completion 2032-04-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of interval cancers | 24-month
  For women at high 2-year risk in the intervention arm interval cancers are defined as cancers diagnosed in the interval between CEM and 12-month mammogram plus in the interval between 12- and 24-month interval. For the remaining women in the trial interval cancers are defined as cancers diagnosed between baseline mammography and 24-month mammography.

SECONDARY OUTCOMES:
Number of recalled women | 24-month
  Information on number of women recalled from screening mammography.

OTHER OUTCOMES:
Number of biopsies | 24-month
  Information on number of biopsies in recalled women.
Breast cancer | 24-month
  Y/N , if yes:date of diagonosis.
Tumor characteristics - Stage | 24-month
  Breast cancer stage 0-4
Tumor characteristics - Multifocality | 24-month
  Unifocal or multifocal
Tumor characteristics - Receptor status | 24-month
  Hormone Receptor Status, to assess the presence of estrogen receptors (ER) and progesterone receptors (PR). HER2 Status, is used to determine whether the cancer cells overexpress the HER2 protein.
Tumor characteristics - Proliferation | 24-month
  Ki-67 Index, provides information about the tumor's proliferative activity.
Cancer worry | 24-month
  Measurement of cancer worry will be done by using answers from the self-reported Cancer Worry Scale (8-item CWS).
  8-item CWS measure cancer worry, score with Likert scale response, four options from min to max cancer worry.
Cancer anxiety | 24-month
  Measurement of cancer anxiety will be done by using answers from the self-reported State Trait Anxiety Inventory (STAI-6).
  STAI-6 measure anxiety. Questions rated on a 4-point Likert scale, options scores from "Not at all" to "Very much" anxiety.
Side effects related to contrast enhanced mammography | 24-month
  The possible side effects related to contrast enhanced mammography and ordinary mammography will be identified using the self-reported Test Morbidity Index.
Cost-effectiveness | 24-month
  Cost-effectiveness will be presented in incremental cost-effectiveness ratio (ICER).
Willingness-to-pay | 24-month
  Willingness-to-pay is defined as the maximum amount that society is willing to pay for each quality adjusted life year (QALY). One quality-adjusted life year (QALY) is equal to 1 year of life in perfect health. Scores range from 1 (perfect health) to 0 (dead).

CONTACTS AND LOCATIONS:
Overall Officials: Per Hall, Professor, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes